CLINICAL TRIAL: NCT02575521
Title: Effect of Propofol-Dexmedetomidine Total Intravenous Anaesthesia on Cerebral Oxygenation and Metabolism During Brain Tumor Resection Compared to Sevoflurane Anaesthesia
Brief Title: Effect of Propofol-Dexmedetomidine on Cerebral Oxygenation and Metabolism During Brain Tumor Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MFM-IRB-14-08-2015
Record Dates: First submitted 2015-10-07; First posted 2015-10-14 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Brain Tumor; Surgery
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol-Dexmedetomidine group (Placebo Comparator): this group is planned to receive intravenous anaesthesia only
  Interventions: Drug: Propofol-Dexmedetomidine group
- Sevoflurane group (Active Comparator): this group is planned to receive sevoflurane/fentanyl anaesthesia
  Interventions: Drug: Sevoflurane group

INTERVENTIONS:
Drug: Propofol-Dexmedetomidine group — Porofol (1.5-2 mg/kg/h) infusion, Dexmedetomidine (0.2-1µg/kg/h) infusion and Fentanyl in repeated doses (50µ) when needed (heart rate or mean arterial blood pressure increase more than 20% of the basal value). Maintenance infusions will start immediately after induction.
  Arms: Propofol-Dexmedetomidine group
Drug: Sevoflurane group — Sevoflurane at a concentration of 2-2.5%., Fentanyl in repeated doses (50µ) when needed (heart rate or mean arterial blood pressure increase more than 20% of the basal value).
  Arms: Sevoflurane group

SUMMARY:
Despite theoretical benefits of intravenous agents, volatile agents remain popular. In a study comparing desflurane, isoflurane, and sevoflurane in a porcine model of intracranial hypertension, at equipotent doses and normocapnia, cerebral blood flow (CBF) and intra-cranial pressure (ICP) were least with sevoflurane.

Propofol is the most commonly used intravenous anesthetic. It has many theoretical advantages by reducing cerebral blood volume (CBV) and ICP and preserving both autoregulation and vascular reactivity. Neurosurgical patients anaesthetized with propofol were found to have lower ICP and higher CPP than those anaesthetized with isoflurane or sevoflurane.

The well known pharmacodynamic advantages of intravenous anesthetics may give this group of drugs superior cerebral effects when compared with inhalation anesthetics.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the cerebral haemodaynamics and global cerebral oxygenation as well as the systemic haemodaynamic changes using dexmedetomidine, propofol and fentanyl as total intravenous anaesthestics (TIVA) in comparison with sevoflurane - fentanyl anesthesia in brain tumor resection.

Indicators of global cerebral oxygenation and haemodynamics will be calculated using jugular bulb and peripheral arterial blood sampling.

* Induction: propofol, 1.5 - 2 mg/kg.
* Muscle Relaxants: atracurium, 0.5 mg/kg with induction and 0.1 mg/kg/20min. for maintenance.
* Cannulation: Arterial cannula: under complete aseptic conditions 20G cannula was inserted into the radial artery of non dominant hand after performing modified Allen's test and local infiltration of 0.5ml xylocaine 2%.

Central venous catheter: A suitable central venous catheter will be inserted into Rt subclavian vein under complete aseptic technique, its correct position will be confirmed with chest X-Ray.

Jugular bulb catheterization: Under strict sterile technique the right internal jugular vein will be cannulated in a retrograde technique with confirmation of the catheter tip position using X-Ray (C- arm). Puncture site will be at the level of cricoid cartilage behind the anterior border of the sternocleido-mastoid muscle.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status III or IV.
* Patients scheduled for elective brain tumor resection

Exclusion Criteria:

* Morbid obese patients.
* Severe or uncompensated cardiovascular diseases.
* Severe or uncompensated renal diseases.
* Severe or uncompensated hepatic diseases.
* Severe or uncompensated endocrinal diseases.
* Pregnancy.
* Postpartum or lactating females.
* Allergy to one of the agents used.
* Severely altered consciousness level.
* Sitting position during surgery.
* Prone position during surgery,

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Arterio-Jugular oxygen content difference | immediately after cannulation (arterial and jugular), every 30 min during surgery and after complete closure of the scalp
Estimated cerebral metabolic rate for O2 (eCMRO2) | immediately after cannulation (arterial and jugular), every 30 min during surgery and after complete closure of the scalp
  eCMRO2=Ca- jO2 x(PaCO2 ∕ 100) Where Ca jO2 is arterio-jugular O2 content difference. PaCO2 is arterial CO2 tension
Cerebral Extraction Rate of O2 (CEO2) | immediately after cannulation (arterial and jugular), every 30 min during surgery and after complete closure of the scalp.
  Calculated as the differences between arterial and jugular bulb O2 saturations, CEO2 = SaO2 - SjvO2
Cerebral Blood Flow equivalent (CBFe) | immediately after cannulation (arterial and jugular), every 30 min during surgery and after complete closure of the scalp
  Which is an index of flow metabolism relationship, calculated as a reciprocal of arterio-jugular O2 content difference. CBFe = 1 ∕CaO2-CjvO.

SECONDARY OUTCOMES:
Heart rate | will be monitored continiously and recorded immediately after intubation, every 30 min during surgery and immediately after closure of the scalp
Blood pressure | will be monitored continiously and recorded immediately after intubation, every 30 min during surgery and immediately after closure of the scalp
End-tidal carbon dioxide tension | will be monitored continiously and recorded immediately after intubation, every 30 min during surgery and immediately after closure of the scalp
Central venous pressure | will be monitored continiously and recorded immediately after intubation, every 30 min during surgery and immediately after closure of the scalp
Postoperative level of sedation | every 5 min for 60 min, after extubation
  all patients will be evaluated using Ramsay sedation scale
Time for first analgesic request from extubation | for 6 hours after surgery
Total analgesics received | for 24 hours after surgery
Intensive care unit stay | for 10 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A. Daif, MD, Principal Investigator — Anaesthesia and Intensive Care Department, College of Medicine, Mansoura University